CLINICAL TRIAL: NCT04278352
Title: Randomized Controlled Trial of Mindfulness-Based Relapse Prevention for Opioid and Alcohol Use Disorders
Brief Title: Mindfulness-Based Relapse Prevention for Opioid and Alcohol Use Disorders
Acronym: MBRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Heidi Zinzow, Professor, Clemson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00084844
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Opioid-use Disorder; Opioid Abuse, in Remission; Alcohol Use Disorder; Alcohol Use Disorder, in Remission
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: Waitlist control design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Relapse Prevention (Experimental): MBRP is a group aftercare program that integrates mindfulness skills training with cognitive-behavioral relapse prevention strategies. The intervention consists of eight weekly two-hour group therapy sessions, delivered by two facilitators with 6-12 people. The experimental group will complete the intervention in weeks 1-8. They will continue treatment as usual for weeks 9-16.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention
- Control (No Intervention): The waitlist control group will not receive the MBRP program during weeks 1-8 and will continue treatment as usual. During weeks 9-16, the control group will receive MBRP.

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — The intervention is a group skills training program that is delivered once weekly for eight weeks. Content focuses on mindfulness and cognitive-behavioral relapse prevention skills, including psychoeducation, experiential exercises, and between session homework assignments.
  Arms: Mindfulness Based Relapse Prevention

SUMMARY:
A randomized controlled trial will examine mindfulness-based relapse prevention (MBRP) program outcomes for 240 individuals who have completed treatment for opioid or alcohol use disorders. MBRP is a group aftercare program that integrates mindfulness skills training with cognitive-behavioral relapse prevention strategies. Primary outcomes will include frequency of opioid/alcohol use, craving, withdrawal, and quality of life. Secondary outcomes include time to first opioid/alcohol use, adherence to medication-assisted treatment plans, perceived stress, posttraumatic stress symptoms, and chronic pain. We will also examine the following potential moderators of intervention outcomes: comorbid diagnoses, life events history, and MBRP intervention adherence. In addition, we will examine the following mediators of intervention outcome: mindfulness skills, emotion regulation skills, executive functioning skills, savoring, and positive and negative affect.

DETAILED DESCRIPTION:
A randomized controlled trial will examine mindfulness-based relapse prevention (MBRP) program outcomes for 240 individuals who have completed treatment for opioid or alcohol use disorders. Participants will be recruited from outpatient medical clinics and substance use recovery centers. They will be assigned to an intervention group (Group 1) or waitlist control (Group 2), completing assessments at baseline, 8, and 16 weeks. Group 1 will receive the intervention in weeks 1-8 and group 2 will receive the intervention in weeks 9-16. MBRP is a group aftercare program that integrates mindfulness skills training with cognitive-behavioral relapse prevention strategies. Primary outcomes will include frequency of opioid/alcohol use, craving, withdrawal, and quality of life. Secondary outcomes include time to first opioid/alcohol use, adherence to medication-assisted treatment plans, perceived stress, posttraumatic stress symptoms, and chronic pain. We will also examine the following potential moderators of intervention outcomes: comorbid diagnoses, life events history, and MBRP intervention adherence. In addition, we will examine the following mediators of intervention outcome: mindfulness skills, emotion regulation skills, executive functioning skills, savoring, and positive and negative affect.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* completed behavioral health treatment for Opioid Use Disorder (OUD) or Alcohol Use Disorder (AUD) within the previous eight weeks
* continues to be followed by a behavioral health provider
* meets DSM-5 criteria for OUD or AUD
* English fluency
* able to attend intervention sessions

Exclusion Criteria

* current psychosis
* dementia
* moderate to severe traumatic brain injury
* pregnancy
* active suicidality
* persistent antisocial behavior
* acute episode of an SUD (past two weeks)
* persistent self-injury requiring clinical management
* already completed or attending a mindfulness-based intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change in frequency of opioid/alcohol use | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Frequency and time to first use will be assessed with both self-timeline follow-back method and collateral timeline follow-back for the past 60 days (Wray et al 2016; Donohue et al., 2004), as well as urine samples.
Change in opioid/alcohol craving | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  We will assess craving with the Penn Alcohol Craving Scale, which will be modified to assess opioid craving for individuals with opioid use disorder (Garland et al., 2014; Flannery, Volpicelli, & Pettinati, 1999). The Penn Scale is a 5 item self-report measure with scores ranging from 0 to 30, with higher scores indicating higher levels of craving.
Change in withdrawal symptoms | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Assessed with The Short Opiate Withdrawal Scale (Gossop, 1990) and the Short Alcohol Withdrawal Scale (Gossop et al., 2002). The Short Opiate Withdrawal Scale and the Short Alcohol Withdrawal Scale are each10 item self-report scales, with scores ranging from 0 to 30, with higher scores indicating more withdrawal symptoms.
Change in quality of life: World Health Organization Quality of Life (WHOQOL)-BREF | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Quality of life will be assessed with the World Health Organization Quality of Life (WHOQOL)-BREF. The WHOQOL-BREF is a 26 item self-report measure that assesses four domains: physical health, psychological, social relationships, and environment. Transformed scores range from 0 to 100 for each of the four domains, with higher scores indicating greater quality of life.

SECONDARY OUTCOMES:
Change in perceived stress | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Perceived stress will be assessed with the Short Form Perceived Stress Scale (PSS-4) (Warttig et al 2013). This scale is 14 items and asks the frequency of feeling stressed on a 0 to 4 scale (total score range of 0-56), with higher scores indicating lower perceived stress.
Change in posttraumatic stress symptoms | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The PTSD Checklist for DSM-5 (PCL-5) will be used to assess PTSD symptoms (Weathers et al, 2013). This scale includes 20 items on a five point scale to assess for PTSD symptom severity. The total score ranges from 0 to 80 with higher scores indicate more severe symptoms.
Change in pain severity: Brief Pain Inventory | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Pain severity will be assessed with the pain severity subscale of the Brief Pain Inventory (Cleeland & Ryan, 1994). The subscale consists of four self-report items (rated 0 to 10), with a total score ranging from 0 to 40. Higher scores indicate higher pain severity.
Change in medication adherence | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Adherence to other medication treatments; 12-item self-report scale, scores range from 12-34, where lower scores indicate better adherence (adherence to medications not given as part of this study) (Kripalani et al. 2009)
Change in mindfulness skills | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The Five Facet Mindfulness Questionnaire (Baer et al, 2006) includes 39 self-report items assessing five dimensions of mindfulness. Items are rated on a 5 point scale ranging from 1 to 5, with total score ranging from 39 to 195. Higher scores indicate greater dispositional tendency to be mindful in daily life (e.g., observing, describing, acting with awareness, nonjudging of inner experience, nonreactivity to inner experiences).
Change in emotion regulation skills | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The Difficulties in Emotion Regulation Scale-Short Form (Kaufman et al., 2016) includes 18 items that assess four areas of emotion regulation: awareness/understanding, acceptance, ability to engage in goal-directed behavior, ability to control impulsive behavior. The items are rated on a 1 (almost never) to 5 (almost always) scale based on frequency of feelings and use of emotion regulation skills, with a total score range of 18-90. Higher scores reflect greater impairments in emotion regulation skills.
Change in executive functioning | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The Executive Function Index has 27-item self-report inventory and assesses five facets of executive functioning (Spinella, 2005); Items rated "how well the following statement describes me" 1 (not at all) to 5 (very much), with a total score range of 27-135, with higher scores indicating higher levels of executive functioning.
Change in Savoring | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The Savoring Beliefs Inventory (Bryant, 2003) is a 24-item self-report instrument with three subscales: anticipating, savoring the moment, and reminiscing. These items are rated on a 1 to 5 scale, half with a negative anchor and half with a positive anchor. Total scores can range from -72 to +72, with higher scores indicating higher levels of savoring.
Change in positive and negative affect | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The Positive and Negative Affect scales assess dispositional dimensions of affect (Watson, Clark, & Tellegen, 1998). Two separate subscales will be used. There are 10 items to evaluate positive affect and 10 items to evaluate negative affect with a range of 10-50 for each scale. Each item is rated according to frequency of feeling a certain way, with higher scores on each scale indicating higher positive or negative affect.

OTHER OUTCOMES:
Satisfaction with Treatment | Assessed at 8 weeks for the experimental group and 16 weeks for the control group.
  The Treatment Satisfaction Survey (Zgierska et al. 2008) is a 5 item self-report measure, with qualitative and quantitative items. The quantitative total scale ranges from 0 to 16, with higher scores indicating greater satisfaction with mindfulness intervention.
Demographics | Assessed at baseline
  Self-report items will assess gender identity, race/ethnicity, family income, health insurance status, educational attainment, marital status, and employment status.
Adverse life event history | Assessed at baseline
  The Adverse Life Events Questionnaire is a 10 item self-report scale assesses adverse events in the first 18 years of life (Felitti, 1998). Total scores range from 0 to 10, with higher scores indicating greater number or adverse events.
Trauma History | Assessed at baseline
  The Life Events Checklist for DSM-5 includes 17 self-report items that assess a number of different types of traumatic events across the lifespan and personal occurrence versus learning about a traumatic event (Weathers et al., 2013). There is no formal scoring protocol, although endorsing 1 or more items indicates lifetime exposure to a traumatic event.
Comorbid Mental Health Conditions | Assessed at baseline
  Current substance use disorders, major depressive disorder, and generalized anxiety disorder diagnoses will be assessed with the respective modules from the Structured Clinical Interview for DSM-5 (First, 2014). Each module includes structured interview questions in "yes/no" response format, with a scoring protocol that indicates whether the participant met criteria for the DSM-5 psychological disorder diagnosis. A categorical outcome will be used (scored "0" for did not meet criteria for the diagnosis, "1" for met criteria for the diagnosis).
Psychological Treatment History | Assessed at baseline
  The Adult Service Use Schedule includes 15 open-ended, self-report items assessing use of psychological services, accessibility, and length of service use (Bower et al., 2000).
Intervention Adherence/Mindfulness Practice Frequency | Assessed at 8 weeks (post-intervention for experimental group), and 16 weeks (follow-up for experimental group, post-intervention for control group)
  Additional mindfulness practices engaged in outside of the study sessions assessed with four self-report items: 'Did you engage in mindfulness meditation in the past month?' (yes = 1, no = 0), 'How many days per week did you engage in mindfulness meditation?' (range = 0-7), 'How long in minutes did you meditate per session of mindfulness meditation?' (range = 0 to unspecified), 'Describe your practice of mindfulness meditation (what exercises/activities/techniques did you practice?). Each quantitative item will be analyzed separately as moderators of intervention outcome and reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shi, Ph.D., Principal Investigator — Clemson University
Locations (3):
- United States (3):
  - Clemson University, Clemson, South Carolina
  - Prisma Health-Upstate Internal Medicine Clinic, Greenville, South Carolina
  - Phoenix Center, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No